CLINICAL TRIAL: NCT00802477
Title: Prospective Randomized Study Comparing Mastectomy Outcomes With Versus Without the Application of Autologous Blood Products to the Surgical Site
Brief Title: Application Of Autologous Blood Products During Modified Radical Mastectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marshall University (Other)
Collaborators: Zimmer Biomet (Industry); Cabell Huntington Hospital (Other)
Responsible Party: Shawn McKinney, MD, Marshall University Joan C. Edwards School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MU9339
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Mastectomy
Keywords: mastectomy; seroma; lymph node dissection
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Application of Autologous Blood Products to surgical site during mastectomy.
  Interventions: Procedure: Application of autologous blood products.
- 2 (Active Comparator): Standard Modified Radical Mastectomy
  Interventions: Procedure: Standard Modified Radical Mastectomy

INTERVENTIONS:
Procedure: Application of autologous blood products. — Autologous blood products (platelet rich and platelet poor plasma) produced by the PlasmaxTM Plus Plasma Concentration System will be applied to the surgical site.
  Arms: 1
Procedure: Standard Modified Radical Mastectomy — Mastectomy per standard procedure without the application of autologous blood products.
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the application of autologous (your own blood) blood products during mastectomy improves wound healing and decreases complications following surgery compared to mastectomy without the use of autologous blood products.

DETAILED DESCRIPTION:
A frequent complication of mastectomy is seroma formation with rates in the literature reported at 3-50%. Although seroma formation can be considered more of a nuisance than a serious complication, the presence of seroma can lead to wound infection, skin flap necrosis, wound dehiscence, nerve injury, and lymphedema in mastectomy patients.Various approaches to reduce seroma formation have included the use of external compression dressings, ultrasound cutting devices, suction drainage systems, and bovine thrombin. Although some of these interventions have demonstrated efficacy, none has gained widespread acceptance. Investigation of alternative interventions during mastectomy procedures that could reduce the rate of postoperative seroma formation, thereby reducing the likelihood of the onset of more serious complications, still has value to the patient and surgeon. The use of autologous blood products (ABP), in particular platelet rich plasma (PRP), has been advocated for numerous indications. As a surgical tool, ABP are typically applied to the surgical site during the latter stages of the procedure in combination with bovine thrombin. The aim of PRP application is to accelerate the healing cascade via application of elevated cytokine concentrations released during platelet degranulation. It is hypothesized that the elevated cytokine levels will elucidate an accelerated healing response of the affected tissue. Preliminary evidence suggests that this expedited healing response correlates with a reduction in postoperative wound complications. Platelet poor plasma, a by-product of PRP processing, has been advocated as providing additional hemostasis. The majority of the literature discussing clinical applications of ABP to date, has been unblinded and nonrandomized. Although useful as demonstrations of the safety of ABP, this current literature does not truly investigate the efficacy of these applications. There is a need for well-designed, well-controlled studies investigating the application of ABP as surgical tools. It is hypothesized that a significant reduction in postoperative complications, in particular seroma formation, will result due to the use of ABP during these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing a modified radical mastectomy, simple mastectomy or axillary lymph node dissection.
2. Patient signature of informed consent form

Exclusion Criteria:

1. Pregnancy
2. < 18 years of age
3. History of anemia (hemoglobin < 11.0)
4. History of any blood disorder, deep vein thrombosis, pulmonary emboli or clotting disorders.
5. Un-cooperative patient or patient with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations
6. Allergy to bovine products
7. History of MRSA in last 12 months
8. Communicable disease or diseases that may limit follow- up (e.g. immunocompromised conditions, hepatitis, active tuberculosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Amount of Drainage during first 7 days postoperative. Drains will be removed during a follow-up visit to be held seven days postoperatively or when drainage is 30-35 ml in a 24 hour period, unless prohibited by complication. | 7 days

SECONDARY OUTCOMES:
The secondary endpoint for this study will be the rate of patients experiencing at least one of the following postoperative wound complications: 1. Seroma Formation 2. Surgical Site Infection | 6 weeks post -op

CONTACTS AND LOCATIONS:
Overall Officials: Shawn McKinney, MD, Principal Investigator — University Physicians and Surgeons, Inc. d/b/a University Oncology Services
Locations (1):
- University Oncology Services at Edwards Comprehensive Cancer Center, Huntington, West Virginia, United States